CLINICAL TRIAL: NCT03709537
Title: Local Organizational Support and Development Networks for Public Mental Health System Workforce With Lived Experience
Brief Title: Supporting the Mental Health Workforce
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Emotional Health Association (Unknown); California Office of Statewide Health Planning and Development (Other)
Responsible Party: Principal Investigator, Louis D. Brown, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSC-SPH-18-0357
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will draw participants from mental health sites where one or more peer supervisors and peer workers are located. These sites will be randomized to either the treatment or standard practice control group. The treatment group will receive the intervention, which consists of a Co-Learning Collaborative, several trainings, and the creation of Implementation Teams. The sites assigned as part of control group will not receive any training or additional technical assistance that is part of the intervention.
Who Masked: Outcomes Assessor
Masking Description: Data collection and analysis will occur without knowledge of participant intervention condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health Peer Workforce Support (Experimental): Sites assigned to this group will engage in Co-Learning Collaborative, several trainings, and the creation of Implementation Teams--all part of the intervention and designed to support their peer workforce.
  Interventions: Behavioral: Mental Health Peer Workforce Support
- Control Group (No Intervention): Sites assigned to this group will continue practice as usual and not receive any additional peer worker training or technical assistance.

INTERVENTIONS:
Behavioral: Mental Health Peer Workforce Support — Supervisors and peer workers will participate in trainings covering effective peer services, trauma-informed effective peer supervision, and responsibilities of peer workers in a supervising relationship. A monthly Supervisors of Peer Workers meeting will support site change efforts. Sites will create an implementation team to work within their site to implement the training received.
  Peer Workers will enroll in a peer mentoring program, where they serve as peer mentors matched with fellow peer mentors. Recovery International and the Los Angeles Department of Mental Health will encourage peer workers to attend Recovery International meetings. Emotional Health Association will refer Peer Workers and their Supervisors in the intervention group to self-help support groups that reduce stress and increase resiliency.
  Arms: Mental Health Peer Workforce Support

SUMMARY:
Emotional Health Association will engage Los Angeles County Department of Mental Health providers that employ peer workers in a training and technical assistance intervention designed to support, increase, and retain an effective peer workforce. This intervention consists of a Co-Learning Collaborative, several training sessions, and the creation of Implementation Teams. Peer workers will also be encouraged to attend Recovery International, an established network of self-help support groups for mental health. Dr. Louis Brown will lead an evaluation of the efficacy of the intervention. This study will inform the use of peer workers as a component of the mental health workforce.

DETAILED DESCRIPTION:
Evaluation of the the intervention with the peer workforce will be conducted through administration of web-based surveys of peer workers and peer supervisors at baseline and follow-up (10 months post-baseline). These two surveys will be administered to peer workers and peer supervisors at sites enrolled in the study. A letter of informational detailing the risks of participation will accompany the survey. Individuals who do not complete the web-based survey will be invited to complete a telephone interview with the same questions. Sites (where one or more peer supervisors and peer workers are located) will be randomized to either the intervention group or standard practice control group. The intervention group will engage in Co-Learning Collaborative, several training sessions, and the creation of Implementation Teams. Peer workers from the intervention group will also be encouraged to attend Recovery International, an established network of self-help support groups for mental health. Analysis of the surveys collected from both study groups will be conducted to assess the efficacy of the intervention and provide Emotional Health Association with a final report.

ELIGIBILITY:
Inclusion Criteria:

* All service providing sites within the Los Angeles Department of Mental Health will be invited to participate in the study. Sites not affiliated with the Los Angeles Department of Mental Health will be allowed to enroll in the study if they express interest but will not be actively recruited.
* Participants must be a peer worker or supervisor of peer workers at a site participating in the study.

Exclusion Criteria:

* Peers who do not receive pay and volunteer for less that 15 hours per week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Peer-supportive organizational climate | 10 months
  Peer-supportive organizational climate will be assessed by a set of 6 likert-scale questions that asks about the participant about his/her organization's administrative leadership and the support they provide.
  1= Strongly Disagree (with positive statement about organization) 7= Strongly Disagree (with positive statement about organization)
Mental Health Stigma | 10 months
  This outcome will be assessed by asking the peer supervisor a set of 15 likert-scale questions about their feelings towards individuals with mental health issues.
  1= Strongly Disagree 5= Strongly Agree
Peer Worker Recovery | 10 months
  This outcome will be assessed by a set of 24 likert scale questions that ask the participants how they feel about themselves and their lives.
  1= Strongly Disagree (with positive statement about self) 5= Strongly Agree (with positive statement about self)

SECONDARY OUTCOMES:
Recovery orientation of services | 10 Months
  This outcome will be measured with 4 questions that ask the peer workers to rate their level of agreement with statements about their organization's treatment of service users (or clients)
  1= Strongly Disagree (with positive statement about services) 7= Strongly Agree (with positive statement about services)
Supervisor's peer support attitudes | 10 Months
  This outcome will be assessed by asking the peer supervisor a set of three likert-scale questions about the importance of peer support for mental health services.
  1=Not important at all 10 =Extremely Important
Supervisor's job satisfaction | 10 Months
  This outcome will be measured using one likert-scale question that asks how satisfied the supervisors are with their job- from 1 (highly unsatisfied) to 5 (very satisfied).
Supervision quality (as rated by peer workers) | 10 Months
  This outcome will be assessed with a set of 7 likert scale questions that ask about the peer worker's experience with their supervisor.
  1= Strongly Disagree (with positive statement about supervisor) 7= Strongly Agree (with positive statement about supervisor)
Peer worker time spent on peer support activities | 10 Months
  This outcome will be measured by asking the peer workers to rate how much time they spend on 9 different support activities on a typical week-- from "None" to "40 hours plus".
Peer worker discrimination experience | 10 Months
  This will be measured with a set of 5 likert scale questions that asks the peer worker about their experience with discrimination due to their mental health.
  1= Strongly Disagree (with statement about negative experience) 5= Strongly Agree (with statement about negative experience)
Supervisor/peer worker relationship (as rated by supervisor) | 10 Months
  This outcome will be measured by a set of 12 likert scale questions from the Supervisory Relationship Measure developed by Pearce et al. 2012.
  1= Strongly Disagree (with positive statement about peer worker) 5= Strongly Agree (with positive statement about peer worker)
Peer worker contributions (as rated by supervisor) | 10 Months
  This outcome will be measured by a set of 12 likert scale questions.
  1= Strongly Disagree 7= Strongly Agree
Peer worker job satisfaction | 10 Months
  This outcome will be measured using one likert-scale question that asks how satisfied the peer workers are with their job- from 1 ("highly unsatisfied") to 5 ("very satisfied").
Peer worker sick leave and disability days | 10 Months
  This outcome will be measured with the following question from the Stapelfeldt et al 2012 instrument:
  "How many sick leave or disability days has _____ had within the last 6 months?"
Peer worker work-related burnout | 10 Months
  This will assesses with a set of 7 likert scale questions that ask the peer worker for the frequency of certain experiences at their job.
  1= Always 5= Never/Almost Never
Peer worker mental health problems | 10 Months
  This outcome will be assessed by a set of 27 likert-scale questions that asks the participant how frequent they have experienced feelings of distress in the past 30 days.
  1= Not all (pertaining to negative statement) 5= Extremely (pertaining to negative statement)
Peer worker social support | 10 Months
  This outcome will be assessed by having the peer workers answer some questions about the people in their environment who provide them with help or support.
  1= Very satisfied (with specific person's support) 6= Very dissatisfied (with specific person's support)
Peer worker stress | 10 Months
  This outcome will be measured by a set of 6 likert scale questions that ask the peer worker to rate the frequency that they have had stressful experiences in the past 30 days.
  1= Never (pertaining to negative statement) 5= Very Often (pertaining to negative statement)

CONTACTS AND LOCATIONS:
Overall Officials: Louis D Brown, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- SHARE! Self-Help and Recovery Exchance, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: No